CLINICAL TRIAL: NCT00579748
Title: Optical Coherence Tomography of the Gastrointestinal Tract
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HS# 2005-4314; Award Number: CA-91717; Proposal Number: 30011
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Barrett's Esophagus With or Without Dysplasia; Patients With Early Esophageal or Gastric Cancer; Patients With Intestinal Metaplasia of the Stomach
Keywords: OCT imaging; Barrett's esophagus
MeSH Terms: conditions — Stomach Neoplasms; Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pinch biopsies blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Optical coherence tomography (OCT) is a non-invasive imaging technique that uses light to create pictures of living tissues and has been successfully used to generate high resolution cross-sectional images of tissue in the human eye and skin. OCT systems are now commercially available for eye and skin use, and several clinical reports on the use of OCT in the gastrointestinal tract have been published as well.

The purpose of this study is to develop a high-speed noninvasive OCT probe which can be placed through an endoscope for the early diagnosis of pre-cancerous and cancerous lesions in the gastrointestinal tract. This is a pilot clinical research study that is designed to advance OCT technology, which may in the future be able to replace or augment endoscopic biopsies.

DETAILED DESCRIPTION:
Protocol Summary The long term objective of the proposed research is to develop a high-speed noninvasive endoscopic functional optical coherence tomography (F-OCT) device using microelectromechanical system (MEMS) technology for early diagnosis of tumors or lesions in gastrointestinal tracts.

Study Design All patients undergoing endoscopy at UCIMC CDDC and who meet eligibility criteria will be candidates for enrollment in the protocol. Signed informed consent will be obtained.

Standard of Care Procedure The patients will undergo the standard of care endoscopy. Endoscopy is performed on a routine basis with conscious sedation or general anesthesia. Digital images and video clips of the areas of interest will be captured in the usual standard of care fashion.

Research Procedure The OCT probe will then be inserted through the biopsy channel of the endoscope into the GI tract lumen and OCT images will be acquired of the lesions just prior to biopsies (research procedure). In addition, OCT images will be taken of the surrounding normal tissue.

Primary Endpoint The OCT images will be correlated to the specific biopsy site and biopsy number.

OCT Device and Probe Optical coherence tomography (OCT) is an emerging imaging modality that uses light to image turbid media such as living tissues, and has been successfully used to generate high resolution (~10 micron) cross-sectional images of tissue microstructure in the human retina and skin. OCT devices are now commercially available for ophthalmic and dermatologic use, and several clinical reports on the use of OCT in the vascular system and aerodigestive tract have been published as well.

The OCT device is an optical imaging instrument that combines a broadband low power near infrared light source (non-laser) with an interferometer to produce cross-sectional optical images of tissue to depths of 1-2 mm. OCT is already used commercially to image the retina and skin. This study focuses on a device designed specifically for the aerodigestive tract. The OCT probe has been designed to fit through the biopsy channel of standard endoscopes. The probes are designed with three different types of mechanism. (1) The first mechanism consists of a fiber optic with a micro lens and prism attached at the end to direct the light to and from the tissue sample. Scanning is achieved by moving the fiber optic along its axis using a linear motor. Longitudinal OCT imaging can be realized with this mechanism. Similar probes are already used in our laryngoscopic OCT study. (2) The second mechanism is achieved by a rotational MEMS motor, on which an angled mirror is attached to direct the light to the side. Rotational imaging can be realized with this mechanism. (3) The third mechanism is based on the silicon MEMS technology. The scanner is created with a polysilicon micromirror driven by high frequency, thick single crystal silicon comb drives. The high speed scanning probe is with large scan angles, excellent optical properties, high precision, and long-term reliability. The overall cross-sectional diameter is approximately 3 mm to be able to fit into the biopsy channel of the endoscope. The OCT device will focus the incident low-coherence light onto the tissue and collect backscattered coherent photons. The endoscopists can then obtain cross sectional optical images of the tissue through arbitrary planes of section.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Barrett's esophagus with or without dysplasia, who are scheduled for surveillance endoscopy with biopsy or endoscopic mucosal resection (EMR).
* Patients with early esophageal or gastric cancer who are undergoing confirmatory endoscopy with biopsy. These cancers must be limited to T1 N0 M0 (tumor invades submucosa with no lymph node involvement and no metastasis) according to the American Joint Committee on Cancer (AJC) Guidelines (1988 or later). Tumors may either be adenocarcinoma or squamous cell cancers. EUS and CT scanning will be required to confirm tumor staging. Tumors must be limited only to the mucosa or submucosa when examined by high frequency c-EUS. Any thickness of tumor lesion is acceptable provided the lesion does not appear to reach the muscularis propria.
* Patients with intestinal metaplasia with or without dysplasia of the stomach who are undergoing endoscopy with biopsy or EMR.
* Patients must be at least 18 years of age. Female patients must not be pregnant (must have a negative serum pregnancy test) or nursing, and must be practicing a medically acceptable form of birth control or be sterile or postmenopausal.
* Patients must sign an informed consent.

Exclusion Criteria:

* Patients with esophageal or gastric cancer, who have tumor extension into the muscularis propria on endoscopic ultrasonography (EUS) (i.e. tumor depth of invasion T2 or greater).
* Patients with esophageal strictures unresponsive to dilation.
* Patients with known contraindications to analgesia or endoscopy.
* Patients with inability to understand or carry out instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve the OCT imaging of patients undergoing endoscopy of the upper digestive tract in the gastrointestinal endoscopy suite in the H. H. Chao Digestive Diseases Center (CDDC) at UC Irvine Medical Center.
  These patients will include: 1) patients with known Barrett's esophagus with or without dysplasia, who are scheduled for surveillance endoscopy with biopsy or endoscopic mucosal resection (EMR) 2) patients with early esophageal or gastric cancer who are undergoing confirmatory endoscopy with biopsy or 3) patients with intestinal metaplasia with or without dysplasia of the stomach who are undergoing endoscopy with biopsy or EMR.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The OCT images will be correlated to the specific biopsy site and biopsy number. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Chang, MD, Principal Investigator — University of California, Irvine; Zhongping Chen, Ph.D., Study Director — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States